CLINICAL TRIAL: NCT05919966
Title: The Association Between Chlorhexidine Bathing Every Other Day and Central Line-Associated Infections in Medical Intensive Care Units: An Observational Cohort Study
Brief Title: The Association Between Chlorhexidine Bathing and Central Line-Associated Infections in Medical Intensive Care Units
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202302031RINC
Record Dates: First submitted 2023-06-13; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-04

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chlorhexidine group: Patients were bathed one day involving the use of wipes soaked in a 2% chlorhexidine gluconate (CHG) solution and the next day using a towel soaked with water and soap during the MICU stays.
  Interventions: Other: Chlorhexidine bathing
- usual care group: Patients were bathed with towels soaked in water and soap on a daily basis during the MICU stays.

INTERVENTIONS:
Other: Chlorhexidine bathing — The procedure involved pouring an entire bottle (200ml) of 2% CHG solution (PBF Biotech, Taipei, Taiwan) onto a pre-packed set of eight single-use cotton wipes before each bathing session. A minimum of six wipes were required to thoroughly cover the entire body, including the bilateral upper and lower extremities, front and back of the trunk, perineum, and buttocks.
  Groups: chlorhexidine group

SUMMARY:
We conducted a retrospective observational cohort study assessing the relationship between regular bathing using 2% CHG wipes every other day and the occurrence of central line-associated infections (CLABSI) in patients within the medical intensive care unit (MICU).

DETAILED DESCRIPTION:
This study defined the post-intervention period as July 1, 2017, to June 30, 2022. During this period, one of the three medical intensive care units (MICUs) in NTUH implemented chlorhexidine gluconate (CHG) bathing as part of their daily care routine (CHG group). This decision was made in response to a higher incidence rate of vancomycin-resistant Enterococcus (VRE) bacteremia observed in that particular MICU during the preceding six months (pre-intervention period: January 1, 2017, to June 30, 2017), compared to the other two MICUs. The remaining two MICUs continued to provide usual care, which involved bathing patients with towels soaked in water and soap on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* all patients who were admitted to the MICU between January 2017 and June 2022

Exclusion Criteria:

* patients aged under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study included all patients aged eighteen years and older who were admitted to the MICU between January 2017 and June 2022, without any exclusions based on specific disease characteristics.
Sampling Method: Probability Sample
Enrollment: 6930 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
central line-associated bloodstream infections | Will be surveyed retrospectively through the study period (January 2017 to June 2022)
  the incidence rate of intensive care unit acquired central line-associated bloodstream infections
multidrug-resistant organisms bacteremia | Will be surveyed retrospectively through the study period (January 2017 to June 2022)
  the incidence of CLABSIs with blood cultures positive for multidrug-resistant organisms

SECONDARY OUTCOMES:
ICU length of stay | Will be surveyed retrospectively through the study period (January 2017 to June 2022)
  the total duration of the patient's ICU stay (days)
hospital length of stay | Will be surveyed retrospectively through the study period (January 2017 to June 2022)
  the total duration of the patient's hospital stay (days)
ICU mortality | Will be surveyed retrospectively through the study period (January 2017 to June 2022)
  whether the patient has died during their stay in the ICU
hospital mortality | Will be surveyed retrospectively through the study period (January 2017 to June 2022)
  whether the patient has died during their stay in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chen Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No